CLINICAL TRIAL: NCT05074446
Title: Stereotype Threat Effect on CPR Performance in Covid-19 Intensive Care Units: A Randomised Controlled Mannequin Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Murat Tümer, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Stereotype Threat on Covid ICU
Record Dates: First submitted 2021-10-10; First posted 2021-10-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Stereotype-threat; COVID-19
Keywords: stereotype threat; COVID-19 Pandemic; non-intensivist physicians; Cardiopulmonary Resuscitation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: It will be a 2x2 between-subject factorial design. Simulation CPR scores will be the dependent variable. Being an intensivist or non-intensivist and stereotype threat will be the independent variables of the study. There will be four groups to be compared: intensivist in the experimental group (1), intensivist in the control group (2), non-intensivist in the experimental group (3), non-intensivist in the control group (4).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- intensivist in the experimental group (Experimental): Stereotype threat manipulation will be performed on the intensivist in the experimental group just before they are taken into the testing room.
  Interventions: Other: stereotype threat manipulation
- intensivist in the control group (No Intervention): The intensivist in the control group will not be given any prior information.
- non-intensivist in the experimental group (Experimental): Stereotype threat manipulation will be performed on the non-intensivist in the experimental group just before they are taken into the testing room.
  Interventions: Other: stereotype threat manipulation
- non-intensivist in the control group (No Intervention): The non-intensivist in the control group will not be given any prior information.

INTERVENTIONS:
Other: stereotype threat manipulation — Stereotype threat is the thought that a person will be negatively evaluated and judged regarding a negative stereotype that belongs to the group to which he/she belongs.
  Stereotype threat manipulation will be performed on the intensivist and non-intensivist participants in the experimental group just before they are taken into the testing room. For manipulation, the following sentences will be said to the participants in the experimental group: "We aim to compare the cardiopulmonary resuscitation performance between intensive care units and other branches." The other participants (Control Group) will not be given any prior information.
  Arms: intensivist in the experimental group; non-intensivist in the experimental group

SUMMARY:
Stereotype threat (ST) is an important issue that has been studied repeatedly in the psychology literature. ST is the thought that a person will be negatively evaluated and judged regarding a negative stereotype that belongs to the group to which he/she belongs. Most people are members of a social group associated with at least one negative stereotype. Therefore, many people in society may be the target of stereotype threat. Previous research has shown that the individual performance of people in groups identified with negative stereotypes, who are exposed to stereotype threat, decreases. The ST may arise when there is an environment in which the skills of the person that may be affected by a stereotype associated with his/her group can be measured, or if this stereotype has become evident.

In Covid-19, there has been a rapid increase in the number of intensive care patients in our country and around the World. Due to this rapid increase, the number of intensivist physicians is insufficient, and non-intensivist physicians from various branches are assigned to intensive care units. In social media and newspaper reports, it was stated that non-intensivist physicians have insufficient knowledge and skills in intubation and in the treatment of lung infection, and the public was asked to take precautions. However, these physicians were expected to treat lung infections and intubate the patients in intensive care units during pandemics. It is unknown to what extent such negative stereotypes, established or already existing, affect the performance of non-intensivist physicians during their appointment to the intensive care units during the pandemic.

As in all other departments, the most basic task expected from doctors in intensive care units is effective basic life support applied for the treatment of cardiopulmonary arrest. Cardiopulmonary resuscitation (CPR) is a basic life support model that is mandatory taught in medical schools. For this reason, it is expected that all doctors, regardless of their specialties, will be able to perform CPR effectively. The use of manikins is quite common in order to standardize CPR training and performance measurement. The aim of this study is to evaluate how non-intensivist physicians assigned to intensive care units during the pandemic are affected by stereotype threat and to investigate the necessary conditions to prevent a possible decrease in performance in these physicians.

ELIGIBILITY:
Inclusion Criteria:

1- To have worked in the Covid-19 intensive care unit during the pandemic

Exclusion Criteria:

1. Not meeting the above criteria
2. Not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Resuscitation (CPR) Performance | During CPR simulation
  Change in CPR scores in the experimental group compared to the control group. Scoring will be done with the "CPR Scoring Scale" we developed. Higher values will indicate more effective CPR.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
İndividual participant data (IPD) will be anonymized to available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: at the end of the study

REFERENCES:
- [Background] Steele CM, Aronson J. Stereotype threat and the intellectual test performance of African Americans. J Pers Soc Psychol. 1995 Nov;69(5):797-811. doi: 10.1037//0022-3514.69.5.797. PMID 7473032
- [Background] Steele, C. M., Spencer, S. J., & Aronson, J. (2002). Contending with group image: The psychology of stereotype and social identity threat. In Advances in experimental social psychology (Vol. 34, pp. 379-440). Academic Press.
- [Background] Steele CM. A threat in the air. How stereotypes shape intellectual identity and performance. Am Psychol. 1997 Jun;52(6):613-29. doi: 10.1037//0003-066x.52.6.613. PMID 9174398
- [Background] Genel Koronavirüs Tablosu. (2021). Retrieved June 22, 2021, from https://covid19.saglik.gov.tr/TR-66935/genel-koronavirus-tablosu.html
- [Background] Baumgaertner, E., & Karlamangla, S. (2020, March 20). Coronavirus outbreak has doctors, nurses bracing for onslaught. Los Angeles Times. https://www.latimes.com/california/story/2020-03-20/coronavirus-doctors-nurses-fears-ventilator-icu-emergency
- [Background] Katipoglu B, Madziala MA, Evrin T, Gawlowski P, Szarpak A, Dabrowska A, Bialka S, Ladny JR, Szarpak L, Konert A, Smereka J. How should we teach cardiopulmonary resuscitation? Randomized multi-center study. Cardiol J. 2021;28(3):439-445. doi: 10.5603/CJ.a2019.0092. Epub 2019 Sep 30. PMID 31565794
- [Background] Ontrup G, Vogel M, Wolf OT, Zahn PK, Kluge A, Hagemann V. Does simulation-based training in medical education need additional stressors? An experimental study. Ergonomics. 2020 Jan;63(1):80-90. doi: 10.1080/00140139.2019.1677948. Epub 2019 Oct 31. PMID 31587619
- [Result] Board, T. [@tim_n_board]. (2020, March 16). #stayhome #covid [Tweet]. Twitter. https://twitter.com/tim_n_board/status/1239499551419047936?s=20

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT05074446/Prot_SAP_002.pdf